CLINICAL TRIAL: NCT03827993
Title: Improving Sexual Health in Gynecologic Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE14818
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine surveillance (No Intervention): Routine surveillance consists of attending gynecologic oncology office visits and being provided with an educational pamphlet discussing common sexual health concerns in gynecologic cancer patients, describing vaginal dilators, moisturizers, and lubrication. Resources for psychosocial counseling, physical therapy, and the sexual health clinic will be provided as well.
  Participants will have follow up at baseline, 3, 6, 9, and 12 months. Baseline visit consists of the initial visit where the Female Sexual Function Index (FSFI) screen was performed. Subsequent follow up visits will consist of FSFI, Female Sexual Distress Scale (FSDS), Kessler 10 surveys, and clinical assessment with Vaginal Assessment Scale and Vulvar Assessment Scale (VAS and VuAS).
- Dedicated sexual health clinic appointment (Experimental): Dedicated sexual health clinic appointment with a physician provider focused on sexual health in this population. This will consist of the provider performing a focused history and physical, who will then determine need for appropriate treatment and management, which may consist of recommendations for medications, psychosocial counseling, physical therapy, and/or dilator use, but are not required.
  The participants will follow up at 3, 6, 9, and 12 months after initial visit, either with the sexual health focused provider or their primary gynecologic oncologist, as determined by the needs of the participant per the provider.
  Interventions: Behavioral: dedicated sexual health clinic appointment

INTERVENTIONS:
Behavioral: dedicated sexual health clinic appointment — Intervention will consist of a dedicated sexual health clinic appointment with a physician provider focused on sexual health in this population. This provider will perform a focused history and physical, and will then determine need for appropriate treatment and management, which may consist of recommendations for medications, psychosocial counseling, physical therapy, and/or dilator use, but are not required.
  Arms: Dedicated sexual health clinic appointment

SUMMARY:
This study seeks to find out if an early intervention of providing directed sexual health education and treatment for gynecologic cancer patients will improve patient outcomes as compared to routine clinic visits.

DETAILED DESCRIPTION:
Participants will be randomly placed to one of two groups. This random placement allows our research study to be more significant when the study team checks the results. In one group, the "control" group, participants will attend their usual clinic visits with their provider every 3 months for a year. At each clinic visit participants will be asked to fill out 3 short surveys (each takes less than 3 minutes). Participants will have a gynecologic exam like they routinely would for cancer surveillance, and confidential notes will be made regarding their exam to assess for improvement or worsening over time.

In the other group, the "intervention" group, participants will attend one focused Sexual Health Clinic visit, where a provider specialized in sexual health for cancer patients will review a focused history and physical, and will provide education, as well as recommend any helpful treatments.

This provider may or may not recommend follow up with her again after this initial visit. Participants will otherwise continue the usual every 3 month clinic visits with their Gynecologic Oncologist for a year. At each clinic visit participants will be asked to fill out 3 short surveys (each takes less than 3 minutes). Participants will have a gynecologic exam like they routinely would for cancer surveillance, and confidential notes will be made regarding their exam to assess for improvement or worsening over time. Participants will not need any additional blood draws or procedures. During their gynecologic exam, a swab will be collected to test participants vaginal pH - a test to see the health of their vaginal flora.

In brief, participants will have their usual 4 clinic visits: one at 3 months, 6 months, 9 months, and 12 months. At each visit, participants will fill out 3 surveys and have a gynecologic exam performed as they usually would, but with a vaginal swab for vaginal pH. This swab will be assessed in the clinic by their provider as the swab will change colors to show pH at the time of exam. This result will be noted in the participants' chart and the swab will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Screening positive for sexual health dysfunction as per baseline FSFI
* Diagnosed with any gynecologic malignancy

It is acceptable to have received treatment prior to or during enrollment, including prior surgery, chemotherapy, radiation, hormonal therapy, or clinical trial.

Exclusion Criteria:

* Unable to speak English
* Patients unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change in sexual dysfunction as measured by FSFI | At 3, 6, 9, and 12 months from start of treatment
  Change in sexual function as measured by FSFI, a 19-question, standardized scale of female sexual function, validated in cancer survivors as compared to start of study.

SECONDARY OUTCOMES:
Change in sexual distress as measured by FSDS | At 3, 6, 9, and 12 months from start of treatment
  Change in sexual distress score as measured by FSDS, a 13-question, validated questionnaire assessing sexually related personal distress in women with female sexual dysfunction. This questionnaire will be used for follow up visits to help assess the level of distress participants are enduring related to their sexual dysfunction.
Change in psychologic distress as measured by Kessler K10 Scale | At 3, 6, 9, and 12 months from start of treatment
  Change in psychologic distress as measured by Kessler K10 Scale, a 10-question, validated questionnaire assessing psychological distress. This survey will be used at follow up visits to help determine baseline psychological distress unrelated to sexual distress for a more global picture of the participants' coping throughout their illness. Scores range from 10 to 50 with higher scores indicating worse distress symptoms.
Change in clinical assessment of vaginal symptoms as measured by VAS | At 3, 6, 9, and 12 months from start of treatment
  Change in vaginal symptoms as measured by VAS, a 4-item validated clinical measure of vaginal health, with scores ranging from 0-12 and higher scores indicating worse symptoms.
Change in clinical assessment of vulvar symptoms as measured by VuAS | At 3, 6, 9, and 12 months from start of treatment
  Change in vulvar symptoms as measured by VAS, a 4-item validated clinical measure of vulvar health with scores ranging from 0-12 and higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ricci, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Sensitive personal information collected regarding sexual health, concern for recruitment of patients with data sharing